CLINICAL TRIAL: NCT04152070
Title: Validation of the Spanish-language Version of the Kihon Checklist to Assess Frailty in Older Adults
Brief Title: Spanish-language Version of the Kihon Checklist
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Trinidad Sentandreu-Mañó, Principal Investigator, University of Valencia
Other Study IDs: H1507116319683
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Frailty
Keywords: Frailty; Spanish; Older adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community-dwelling older adults: Community-dwelling older adults living in the Valencia region (Spain).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There was no intervention to be administered, only collection of data through various tests and questionnaires.

SUMMARY:
The purpose of this cross-sectional study is to validate the Spanish version of the Kihon Checklist for screening frailty in Spanish community-dwelling older adults.

DETAILED DESCRIPTION:
In order to identify individuals at risk for frailty, a wide variety of assessment tools have been developed in recent years. Nevertheless, there is still a lack of a gold standard method to be used. Therefore, simple, reliable, and valid instruments are still needed for both research and clinical purposes. The Kihon Checklist is a multidimensional tool widely used in Japan and in other countries, but an exhaustive validity in Spanish population has not been yet established.

The main objective is to validate the Spanish version of the Kihon Checklist for screening frailty in Spanish community-dwelling older adults, and as a secondary objective, to study and to compare different scales of frailty in the Spanish population, and to study their associations.

To cope with the objectives of the present study, a cross-sectional study was conducted. To this purpose, data were collected through various tests and questionnaires about: frailty; clinical, demographic and anthropometric characteristics; physical assessment; functional status; cognitive function; health-related quality of life; depressive mood; and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Community-dwelling older adults

Exclusion Criteria:

* Barthel Index < 85 points considering as disabled
* Mini-Mental State Examination < 18 points
* Acute disease
* Unstable chronic disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community-dwelling older adults living in the Valencia region.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Frailty: The Kihon Checklist | The cohort group was assessed in one day visit.
  The Kihon Checklist is a self-reporting survey used for screening frail older adults. It consists of 25 yes/no questions divided into 7 domains: activities of daily living, physical strength, nutrition, eating, socialization, memory, and depressive mood. Higher scores indicate a higher risk of requiring support. A total score ≥ 7 points indicates general frailty (Sewo Sampaio 2016). The Spanish Kihon version used for validation in this study was translated by Maseda et al. (2017).
Frailty: Fried's Frailty Phenotype | The cohort group was assessed in one day visit.
  Fried's Frailty Phenotype proposed in the Cardiovascular Health Study (Fried 2001) consists of 5 criteria: unintentional weight loss, exhaustion, low physical activity, reduced grip strength, and reduced gait speed. It has a total score ranging from 0 to 5. A frail person is who scores 3 to 5; prefrail when scores 1 to 2, and robust when scores 0.
Frailty: The Edmonton Frailty Scale | The cohort group was assessed in one day visit.
  The Edmonton Frailty Scale (Rolfson 2006) evaluates 9 domains of frailty: cognition, general health status, functional independence, social support, medication usage, nutrition, mood, continence, and functional performance. It has a total score ranging from 0 to 17, with higher scores representing greater frailty severity.
Frailty: The Frail Scale | The cohort group was assessed in one day visit.
  Frailty measured by the Frail Scale (Masanes et al., 2012). It has a total score of 5 points. The more score the more frailty. Participants are considered frail individuals with scores 3 to 5; prefrail with scores 1 to 2, and robust with scores of 0.
Frailty: The Tilburg Frailty Indicator | The cohort group was assessed in one day visit.
  The Tilburg Frailty Indicator (Gobbens et al., 2010) is a self-reported questionnaire of 15 items addressing physical, psychological and social domains. The total score of the Tilburg scale can range from 0 to 15. Higher scores indicate more frailty.

SECONDARY OUTCOMES:
Handgrip strength | The cohort group was assessed in one day visit.
  Muscle strength was measured by the isometric handgrip strength (Cruz-Jentoft et al., 2010).
Knee extension strength | The cohort group was assessed in one day visit.
  Muscle strength was measured by the isometric knee extension (Andrews et al., 1996).
Elbow flexion strength | The cohort group was assessed in one day visit.
  Muscle strength measured by the isometric elbow flexion (Andrews et al., 1996).
Muscle mass | The cohort group was assessed in one day visit.
  Muscle mass estimated by Bioimpedance analysis (BIA) (Bahat et al., 2016).
Gait speed | The cohort group was assessed in one day visit.
  Gait speed was recorded using a 4-meter walking test (Working Group on Functional Outcome Measures for Clinical Trials, 2008).
Modified Baecke Questionnaire | The cohort group will be assessed in one day visit.
  Physical condition was measured by the Modified Baecke Questionnaire (Vilaró et al., 2007). The Modified Baecke Questionnaire results in a score to classify people as high, moderate, or low in daily physical activity, based on tertiles.
The Short Physical Performance Battery | The cohort group was assessed in one day visit.
  Physical performance was measured by the Short Physical Performance Battery (Guralnik, 1994). This measurement consists of walking 4m, a balance test with 3 levels (tandem, semi-tandem and stand up on one foot) and sit up and reach 5 times as fast as possible. Summary scores range from 0-12, and higher scores denote higher physical performance.
Barthel Index | The cohort group was assessed in one day visit.
  Functional independence was measured by the Barthel Index. It has a total score ranging from 0 to 100, where 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
Lawton and Brody Questionnaire | The cohort group will be assessed in one day visit.
  Functional independence was measured by the Lawton and Brody Questionnaire (Lawton and Brody, 1969). Instrumental activities of daily living assess the ability to use the telephone, to shop, to use transport, to cook, to do housework, to take medication, and to handle finances. It has a total score ranging from 0 to 8, 0 indicates total dependence and the maximum score indicates total independence.
Mini-Mental State Examination | The cohort group was assessed in one day visit.
  Cognitive function was measured by the Spanish version of the Mini-Mental State Examination (Lobo et al., 1999). Summary scores range from 0 to 35, and higher scores denote higher cognitive function.
Short Form Health Survey SF-8 | The cohort group was assessed in one day visit.
  Health-related quality of life was measured by SF-8 (Tomás et al., 2017). Summary scores range from 8 to 40, and higher scores denote a higher health-related quality of life.
Depressive symptoms CES-D short form (CESD-7) | The cohort group was assessed in one day visit.
  Depressive mood was measured by CESD-7 (Herrero y Gracia, 2007). Summary scores range from 0 to 21, and lower scores denote depressive mood.
Mini Nutritional Assessment-Short Form (MNA-SF) | The cohort group was assessed in one day visit.
  Nutritional status was measured by MNA-SF (Rubenstein et al., 2001). Summary scores range from 0 to 14, and higher scores denote better nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: Trinidad Sentandreu Mañó, PT, PhD, Principal Investigator — University of Valencia; Jose M. Tomas, PhD, Study Chair — University of Valencia; J. Ricardo Salom Terrádez, PhD, Study Chair — Doctor Peset University Hospital, Valencia, Spain; Mercè Balasch i Bernat, PT, PhD, Study Chair — University of Valencia; Natalia Cezón Serrano, PT, Study Chair — University of Valencia; Maria A Cebrià i Iranzo, PT, PhD, Study Chair — University of Valencia; Maria A Tortosa Chuliá, PhD, Study Chair — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

REFERENCES:
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Bahat G, Tufan A, Kilic C, Karan MA, Cruz-Jentoft AJ. Methodological issues in determination of low muscle mass reference cut-off values: Reply to Comment on "Cut-off points to identify sarcopenia according to European Working Group on Sarcopenia in Older People (EWGSOP) definition". Clin Nutr. 2017 Jun;36(3):903-904. doi: 10.1016/j.clnu.2017.02.023. Epub 2017 Mar 11. No abstract available. PMID 28336166
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Herrero J, Gracia E. A [Brief Measure of Depressive Symptomatology (CESD-7)]. Salud Ment 2007;30(5):40-46.
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Lobo A, Saz P, Marcos G, Dia JL, de la Camara C, Ventura T, Morales Asin F, Fernando Pascual L, Montanes JA, Aznar S. [Revalidation and standardization of the cognition mini-exam (first Spanish version of the Mini-Mental Status Examination) in the general geriatric population]. Med Clin (Barc). 1999 Jun 5;112(20):767-74. Spanish. PMID 10422057
- [Background] Masanes F, Culla A, Navarro-Gonzalez M, Navarro-Lopez M, Sacanella E, Torres B, Lopez-Soto A. Prevalence of sarcopenia in healthy community-dwelling elderly in an urban area of Barcelona (Spain). J Nutr Health Aging. 2012 Feb;16(2):184-7. doi: 10.1007/s12603-011-0108-3. PMID 22323356
- [Background] Maseda A, Lorenzo-Lopez L, Lopez-Lopez R, Arai H, Millan-Calenti JC. Spanish translation of the Kihon Checklist (frailty index). Geriatr Gerontol Int. 2017 Mar;17(3):515-517. doi: 10.1111/ggi.12892. No abstract available. PMID 28345232
- [Background] Rolfson DB, Majumdar SR, Tsuyuki RT, Tahir A, Rockwood K. Validity and reliability of the Edmonton Frail Scale. Age Ageing. 2006 Sep;35(5):526-9. doi: 10.1093/ageing/afl041. Epub 2006 Jun 6. No abstract available. PMID 16757522
- [Background] Rubenstein LZ, Harker JO, Salva A, Guigoz Y, Vellas B. Screening for undernutrition in geriatric practice: developing the short-form mini-nutritional assessment (MNA-SF). J Gerontol A Biol Sci Med Sci. 2001 Jun;56(6):M366-72. doi: 10.1093/gerona/56.6.m366. PMID 11382797
- [Background] Sewo Sampaio PY, Sampaio RA, Yamada M, Arai H. Systematic review of the Kihon Checklist: Is it a reliable assessment of frailty? Geriatr Gerontol Int. 2016 Aug;16(8):893-902. doi: 10.1111/ggi.12833. PMID 27444395
- [Background] Tomas JM, Galiana L, Fernandez I. The SF-8 Spanish Version for Health-Related Quality of Life Assessment: Psychometric Study with IRT and CFA Models. Span J Psychol. 2018 Mar 22;21:E1. doi: 10.1017/sjp.2018.4. PMID 29562950
- [Background] Vilaro J, Gimeno E, Sanchez Ferez N, Hernando C, Diaz I, Ferrerc M, Roca J, Alonso J. [Daily living activity in chronic obstructive pulmonary disease: validation of the Spanish version and comparative analysis of 2 questionnaires]. Med Clin (Barc). 2007 Sep 15;129(9):326-32. doi: 10.1157/13109543. Spanish. PMID 17910846
- [Background] Working Group on Functional Outcome Measures for Clinical Trials. Functional outcomes for clinical trials in frail older persons: time to be moving. J Gerontol A Biol Sci Med Sci. 2008 Feb;63(2):160-4. doi: 10.1093/gerona/63.2.160. No abstract available. PMID 18314451